CLINICAL TRIAL: NCT05754463
Title: The Effect Of Plyometric Training On Balance And Proprioception
Brief Title: The Effect Of Plyometric Training On Balance And Proprioception In Different Branches Athletes
Acronym: Plyometric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mustafa gulsen (Other)
Collaborators: Okan University (Other)
Responsible Party: Sponsor-Investigator, mustafa gulsen, assocc.prof.dr., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 40
Record Dates: First submitted 2023-02-07; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Athlete Foot
Keywords: Plyometrics; Balance; Proprioception
MeSH Terms: conditions — Tinea Pedis | interventions — Proprioception

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- athletes (Experimental): Plyometric training was applied to the athletes (Group 1) (n=27) participating in our study, 2 days a week for 6 weeks, after 20 minutes of warming up and stretching movements before each training. Sociodemographic characteristics of the athletes were recorded. Dynamic balance test was applied with Y balance test and static balance was applied with strok balance test before and after plyometric training. Proprioception assessment was applied with kinematic angle reproduction test before and after plyometric training.
  Interventions: Other: The effect of plyometric training on balance and proprioception in athletes in different branches
- karate (Active Comparator): Plyometric training was applied to the karate practitioners (Group 2) (n=27) participating in our study, 2 days a week for 6 weeks, after 20 minutes of warming up and stretching movements before each training. Sociodemographic characteristics of the athletes were recorded. Dynamic balance test was applied with Y balance test and static balance was applied with strok balance test before and after plyometric training. Proprioception assessment was applied with kinematic angle reproduction test before and after plyometric training.
  Interventions: Other: The effect of plyometric training on balance and proprioception in athletes in different branches

INTERVENTIONS:
Other: The effect of plyometric training on balance and proprioception in athletes in different branches — Investigating the effect of plyometric training on balance and proprioception in athletes in different branches

SUMMARY:
The aim of this study is to investigate the effect of plyometric training on balance and proprioception in athletes in different branches.

54 athletes participated in the study. Two groups were included as 27 athletics and 27 karate groups. Plyometric training was applied to the athletes participating in our study, 2 days a week for 6 weeks, after 20 minutes of warming up and stretching movements before each training. Sociodemographic characteristics of the athletes were recorded. Dynamic balance Y balance test and static balance Stroke balance test; sense of proprioception was evaluated with Angle reproduction test.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed athlete in the province of Tokat
* Being an athlete who trains regularly
* To be healthy, between the ages of 12 and 18
* Volunteering to work.

Exclusion Criteria:

* Presence of any disturbance that may affect balance and balance reactions,
* Musculoskeletal injury in the last 6 months,
* Presence of previous musculoskeletal surgery,
* Pregnancy,
* Having an acute or chronic illness or injury that will limit performance in training or a match,
* Calcification or other bone and joint problems,
* Using cigarettes, alcohol, and drugs that affect balance.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Plyometric training | 2 days a week for 6 weeks
  The individuals included in our study were divided into two groups by a simple randomization method. Plyometric training was applied to the both groups (athletes and karate practitoners).
Y balance Test | 6 weeks
  It is used to dynamically measure balance. This test includes extensions in the anterior, posterolateral, and posteromedial directions. .
Stroke Balance Test | 6 weeks
  The athlete warms up for 10 minutes. The athlete stands comfortably on both feet, his hands are on his hips. The athlete raises the right leg and places the sole of the right foot on the edge of the left kneecap. The tester gives the command "GO", starts the stopwatch, and the athlete raises the heel of the left foot and stands on the toes.
Proprioception assessment (Eyes-closed kinematic angle reproduction test) | 6 weeks
  Participants in this test were asked to stand on one leg. The goniometer support point is placed lateral to the knee joint, one side parallel to the trochanter major line, and the other side along the lateral malleola line with the knee extended. In order to get results, the goniometer is fixed. The participant is asked to bring the knee from extension to flexion and stop the knee at a target angle of 30 degrees of flexion at a very low speed (about 10 degrees per second). The participant is asked to remain in this position for 4 seconds and then to extend the knee. The participant is asked to close their eyes and flex the knee to a target degree. In this way, the degree of deviation of the participant is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Gulsen, Study Director — Baskent University
Locations (1):
- The Effect of Plyometric Training on Balance and Proprioception in Different Branches Athletes, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes